CLINICAL TRIAL: NCT03738111
Title: A Phase 1 Dose-Escalation and Pharmacokinetic Study of TG02 Citrate in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of TG02 Citrate in Patients With Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's commercial decision
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: China Oncology Focus Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COF-HK-001
Record Dates: First submitted 2018-11-01; First posted 2018-11-13 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TG02 Citrate (Experimental): TG02 citrate capsules given orally.
  Interventions: Drug: TG02 Citrate

INTERVENTIONS:
Drug: TG02 Citrate — TG02 citrate capsules

SUMMARY:
This is a single-centre, open-label, dose escalation, Phase 1 study. The primary objective is to determine the highest dose of TG02 citrate that can safely be given to patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at screening;
2. Life expectancy ≥ 3 months;
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1;
4. Subjects must have histologically confirmed locally advanced or metastatic hepatocellular carcinoma (HCC) and have tumor that is refractory to or progressive after sorafenib treatment. Or the subjects are intolerable to sorafenib.
5. Prior local therapy to tumor (e.g. surgery, radiofrequency ablation, percutaneous ethanol injection, chemo-embolization, radiotherapy) is allowed provided that there is a target lesion not subjected to local therapy and/or disease progression has been documented in the target lesion subjected to local therapy. The treatment must be completed at least 4 weeks and patient has recovered from all the acute toxicities of that treatment.
6. At least 28 days, or at least 5 half-lives (whichever is shorter), since last systemic therapy (i.e., chemotherapy, targeted therapy, immunotherapy) before the first dosing of TG02, and have recovered from any clinically significant toxicity associated with such treatment;
7. HCC subjects must be of Child-Pugh class A (not amenable to or refractory to locoregional therapy). Subjects with HCC associated with hepatitis B virus must be receiving adequate antiviral therapy.
8. Must have at least 1 measurable lesion per RECIST 1.1 and evidence of disease progression since the last anti-tumor therapy.
9. Adequate hematologic, renal and hepatic function:

   White Blood Cells ≥2000/uL Neutrophils ≥1500/uL Platelets ≥75,000/uL Hemoglobin ≥9.0g/dL (may have been transfused) Creatinine ≤2mg/dL Aspartate Aminotransferase (AST) <5 x upper limit of normal (ULN) alanine aminotransferase (ALT) <5 x upper limit of normal (ULN) Bilirubin ≤2 x ULN (except subjects with Gilbert's syndrome, who must have total bilirubin <3.0mg/dL) INR ≤1.5
10. Persistent clinically significant toxicities from prior chemotherapy must be ≤ grade 1.
11. Ability to take oral medicine.
12. Negative urine pregnancy test at the time of first dose for women of child bearing potential (WOCBP). For men and WOCBP, adequate contraception must be used throughout the study. For this study, acceptable methods of contraception include a reliable intrauterine device or a spermicide in combination with a barrier method. Hormonal forms of birth control (oral, implantable, or injectable) may only be used if combined with a barrier method.
13. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.

Exclusion Criteria:

1. Past liver transplantation.
2. Uncontrollable hepatic encephalopathy or ascites.
3. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, and myocardial infarction within 6 months prior to first dose.
4. Screening ECG with a prolonged QTc interval (males: >450ms; females: >470ms) as calculated by the Fridericia correction formula despite balancing of electrolytes and/or discontinuing any drugs known to prolong QTc interval.
5. Concurrent severe or uncontrolled medical disease (e.g., active systemic infection, diabetes, hypertension, coronary artery disease) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
6. Symptomatic CNS or brain metastases.
7. Psychiatric illness/social situations that would limit compliance with study requirements.
8. Prior or second malignancy, except non-melanoma skin cancer, completed resected cervical or prostate cancer (with prostate-specific antigen (PSA) of less than or equal to 0.1ng/ml), or other cancer for which the subjects has received curative therapy at least 3 years prior to study entry.
9. Patient with pleural effusions requiring thoracentesis or ascites requiring paracentesis.
10. Acute hepatitis.
11. The subject is receiving an investigational drug, has an investigational device in place or has participated in an investigational drug or device study within 30 days prior to screening.
12. Pregnant or nursing.
13. History of drug abuse and taking drugs (such as marijuana, cocaine, opiates, benzodiazepines, amphetamines, barbiturates).
14. History of addicted to alcohol within 6 months before the study which defines as an average weekly intake of greater than 14 units (one unit=17.7ml ethanol, which is equivalent to 357ml beer with 5% alcohol content or 44ml spirits with 40% alcohol content or 147ml wine with 12% alcohol content).
15. Subjects who, in the opinion of the investigators, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  To assess the number of patients with dose-limiting toxicities (DLT) and the dose of TG02 citrate that can be safely given to patients with advanced hepatocellular carcinoma.

SECONDARY OUTCOMES:
Adverse Event | up to 12 months
  All adverse events will be graded according to NCI-CTCAE, Version 4
Objective Response Rate, with respect to RECIST version 1.1 | Up to 12 months
  Proportion of patients, whose best overall response is either Complete Response or Partial Response, confirmed at least 4 weeks after initial documentation.
Progression Free Survival | At progression, up to 12 months
Overall Survival | At death, up to 12 months

OTHER OUTCOMES:
Molecular Marker | At baseline
  Correlation of molecular marker, c-MYC, with measures of clinical benefit.

IPD SHARING:
Plan to Share IPD: No